CLINICAL TRIAL: NCT01997788
Title: The Efficacy of Intrathecal Morphine in Patients Undergoing Open Nephrectomy
Brief Title: The Intrathecal Morphine for Nephrectomy
Acronym: EMPON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Deok Man Hong, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITMPKidney
Record Dates: First submitted 2013-09-10; First posted 2013-11-28 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Renal Cell Carcinoma
Keywords: Injection, Spinal; Morphine; Analgesia; Patient-Controlled; Pain; Postoperative; Combined Modality Therapy; Nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell; Agnosia; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The ITM group (Experimental): The postoperative pain management includes both the intrathecal morphine injection and the intravenous patient-controlled analgesia. Demerol on demand will be injected intravenously.
  Interventions: Drug: The intrathecal morphine injection; Drug: The intravenous patient-controlled analgesia; Drug: Demerol on demand
- The IV-PCA group (Placebo Comparator): The postoperative pain management includes only the intravenous patient-controlled analgesia. Demerol on demand will be injected intravenously.
  Interventions: Drug: The intravenous patient-controlled analgesia; Drug: Demerol on demand

INTERVENTIONS:
Drug: The intrathecal morphine injection — A single injection of morphine intrathecally
  Arms: The ITM group
Drug: The intravenous patient-controlled analgesia — The intravenous injection of morphine using the patient-controlled analgesia machine
Drug: Demerol on demand — Demerol 25 mg intravenously when pain scores more than 5.

SUMMARY:
To evaluate the efficacy and the safety of the intrathecal morphine injection in the open nephrectomy.

DETAILED DESCRIPTION:
The open nephrectomy is the treatment of choice for live donor kidney transplantation and renal cell carcinoma. The incision for the nephrectomy causes severe postoperative pain. A single dose of intrathecal morphine(ITM) has been used for the postoperative pain of prostatectomy, transurethral resection of the prostate and hepatectomy. The effect of ITM for open nephrectomy has not been studied. Therefore, this prospective, randomized study will evaluate the efficacy and safety of a single 50 mcg dose of ITM added to intravenous patient controlled analgesia(IV-PCA), comparing to IV-PCA alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for the open nephrectomy

Exclusion Criteria:

* Patients with renal insufficiency
* Patients with coagulopathy
* History of any neurologic disorder
* History of recent infection in 2 weeks
* History of drug abuse
* Patients who cannot understand the usage of th intravenous patient-controlled analgesia
* Patients using opioids due to the chronic pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The evaluation of pain at 24 hours after surgery | at postoperatively 24 hours
  The doctor blinded to the investigation will visit patients. The pain will be assessed at rest and at coughing using visual analogue scale.

SECONDARY OUTCOMES:
The consumption of analgesics | at postoperatively 24 hours
  The total amount of opioids (IV morphine) used for 24 hours after surgery will be recorded and compared.
The consumption of intraoperative opioids | From the induction of anesthesia till the emergence of anesthesia, an expected average of 4 hours
  The total amount of intraoperative opioids (IV remifentanil) will be recorded and compared.
The side effects of opioids after surgery | During 72 hours after the end of surgery
  Any side effects of opioids including nausea, vomiting, dizziness, sedation, headache, pruritus and respiratory depression will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Deok-Man Hong, PhD, Study Director — Seoul National University of Hospital
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea